CLINICAL TRIAL: NCT03844126
Title: Adolescents With Type 1 Diabetes Who Attend Pre-transition Classes, Are Better Prepared to Transition Their Care From Pediatric to Adult Providers
Brief Title: Transition of Diabetes Care From Pediatric to Adult Healthcare Providers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kanthi Bangalore Krishna, Assistant Professor, Department of Pediatrics, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY0007974
Record Dates: First submitted 2018-06-11; First posted 2019-02-18 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Transition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients attending the classes (Experimental): The patients attending the transition classes will receive a survey to assess transition preparedness before and after attending the class.
  Interventions: Other: Transition classes

INTERVENTIONS:
Other: Transition classes — 90 minutes spent with patients and their families (separately) to review the changes and challenges associated with healthcare transition and help alleviate some of the barriers traditionally associated with this process.

SUMMARY:
A dedicated pre-transition class, as proposed in this study, could help facilitate a smooth transition between pediatric and adult diabetes care. The innovation in this study is that these classes are an opportunity for the patients and their families to meet with the Adult Diabetes Team consisting of a diabetologist, RD and CDE, prior to the transition of care. Having met them would then increase the likelihood of compliance with the Adult clinic visits.

ELIGIBILITY:
Inclusion Criteria:

Adolescents with Type 1 Diabetes

Exclusion Criteria:

Not wanting to participate in the classes

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Transition preparedness | 1 month
  Patients with be given the modified TRAQ questionnaire before and after the program. A team consisting of an adult diabetes provider, diabetes nurse educator and dietitian will meet in small groups with adolescents between ages 16-18 years to provide them with 'adult specific' goals and discuss various topics like college preparedness, expectations from adult providers, potential changes in dynamics of diabetes management etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kanthi Bangalore Krishna, MD, Principal Investigator — PSHMC
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided